CLINICAL TRIAL: NCT04387838
Title: Study of the SARS-COV-2 (COVID-19) Serological Profile of an Army Training Hospital Staff
Acronym: SEROSARSCOV
Status: Completed | Type: Observational
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-COVID19-10; 2020-A01028-31 (Other: IDRCB)
Record Dates: First submitted 2020-05-13; First posted 2020-05-14 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Sars-CoV2
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Anti-SARS-CoV2 serological status: At Day 0, a blood sample is collected by venipuncture and a questionnaire is being filled. The anti-SARS-CoV2 serological status is measured by automated microplate ELISA technique on the EVOLIS analyzer (Biorad®), using reagent kits from EUROIMMUN France.
  For individuals who are anti-SARS-CoV2 seronegative, the same intervention is made at Day 30 and D60.
  For the individuals who are anti-SARS-CoV2 seropositive, the study follow-up is stopped.
  Interventions: Diagnostic Test: Anti-SARS-CoV2 Serology; Other: Questionnaire

INTERVENTIONS:
Diagnostic Test: Anti-SARS-CoV2 Serology — A blood sample is collected by venipuncture at Day 0, Day 30 and Day 60. The anti-SARS-CoV2 serological status is measured by automated microplate ELISA technique on the EVOLIS analyzer (Biorad®), using reagent kits from EUROIMMUN France.
Other: Questionnaire — Data concerning personal exposure factors are collected in a questionnaire:
  * Socio-demographic factors: sex, age
  * Professional factors: Employment (type, pace, reception, service, care practices), wearing of personal protective equipment (type of equipment, frequency of use) and type of hospital
  * Non-professional factors: Contact with infected individuals, carrying of professional equipment and compliance with barrier measures

SUMMARY:
Emerging in China in December 2019, Covid-19, whose pathogen is SARS-Cov-2, was declared a global pandemic in March 2020. The clinical presentation is highly variable, ranging from asymptomatic forms to acute respiratory distress and even death. Transmission occurs through droplets, with a R0 of approximately 3.

Rapidly, population protection measures were put in place by governments, including the confinement of all persons whose functions were not considered essential and the closure of educational institutions.

Health care institutions are places at risk of Covid-19 transmission and hospital staff are particularly exposed, either through direct contact with patients, contact with exposed persons or through the environment. In order to protect personnel, hygiene measures were immediately recalled and reinforced.

This study is aimed at evaluating the incidence rate of anti-SARS-Cov2 seroconversion over 2 months among hospital staff, without any supposed anti-Covid treatment 19.

ELIGIBILITY:
Inclusion Criteria:

* Army Training Hospital staff

Exclusion Criteria:

* Individuals who have already been confirmed Covid-19 positive
* Individuals taking preventive anti-Covid-19 therapy or considering participating in anti-Covid-19 therapy study
* Individuals on hydroxychloroquine
* Pregnant or breastfeeding women
* Non-permanent staff during the study period
* Individuals identified for a detachment outside the metropole during the study period

Ages: 18 Years to 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population is composed of army training hospital staff who have not already been confirmed Covid-19 positive and who are not taking any treatment relative with Covid-19.
Sampling Method: Non-Probability Sample
Enrollment: 845 (Actual)
Dates: Start 2020-05-14 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2020-08-15 (Actual)

PRIMARY OUTCOMES:
Anti-SARS-Cov2 seroconversion between Day 0 and Day 60. | From Day 0 to Day 60
  Change of Anti-SARS-Cov2 serological status between Day 0 and Day 60, measured in blood sample.
Anti-SARS-Cov2 seroconversion between Day 0 and Day 30. | From Day 0 to Day 30
  Change of Anti-SARS-Cov2 serological status between Day 0 and Day 30, measured in blood sample.
Anti-SARS-Cov2 seroconversion between Day 30 and Day 60. | From Day 30 to Day 60
  Change of Anti-SARS-Cov2 serological status between Day 30 and Day 60, measured in blood sample.

SECONDARY OUTCOMES:
Anti-SARS-Cov2 seroprevalence at Day 0. | Day 0
  Anti-SARS-Cov2 seroprevalence measured in blood sample collected at Day 0.
Correlation between seroconversion and socio-demographic factors - sex | Day 60
  Correlation between seroconversion (measured in blood sample) at Day 60 and sex
Correlation between seroconversion and socio-demographic factors - age | Day 60
  Correlation between seroconversion (measured in blood sample) at Day 60 and age
Correlation between seroconversion and professional factors - job type | Day 60
  Correlation between seroconversion (measured in blood sample) at Day 60 and job type (nurse, physician, etc.)
Correlation between seroconversion and professional factors - personal protective equipment type | Day 60
  Correlation between seroconversion (measured in blood sample) at Day 60 and personal protective equipment type
Correlation between seroconversion and non-professional factors - contact with infected individuals | Day 60
  Correlation between seroconversion (measured in blood sample) at Day 60 and contact with infected individuals
Correlation between seroconversion and non-professional factors - wearing of professional equipment | Day 60
  Correlation between seroconversion (measured in blood sample) at Day 60 and wearing of professional equipment
Correlation between seroconversion and non-professional factors - respect of barrier gestures | Day 60
  Correlation between seroconversion (measured in blood sample) at Day 60 and respect of barrier gestures

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital d'Instuction des Armées Sainte-Anne, Toulon
  - Hôpital d'Instruction des Armées Robert Picqué, Villenave-d'Ornon